CLINICAL TRIAL: NCT05570162
Title: Clinical Efficacy of a Diabetes Educational Program to Improve Intermittently Continuous Glucose Monitoring (Flash) Adherence in Type 1 Diabetes Patients
Brief Title: Clinical Efficacy of a Diabetes Educational Program to Improve Flash Adherence in Type 1 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Castilla-La Mancha Health Service (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-558
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: 30 minutes diabetes educational program:
  * 10-minute talk about Flash measurements and importance of diabetes control.
  * 10-minute practic exercises with Flash values and tendencies.
  * 10-minute talk about recomendations for increasing daily Flash scanning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Low Flash adherence (Experimental): Adult (>18 yrs old) type 1 diabetes patients with 4 or less daily Flash scans
  Interventions: Other: Diabetes educational program

INTERVENTIONS:
Other: Diabetes educational program — 30-minute long diabetes educational program

SUMMARY:
Prospective observational study to analyse the clinical effectiveness of a diabetes educational program to improve intermittently continuous glucose monitoring (iCGM) adherence in adult type 1 diabetes (T1D) patients

DETAILED DESCRIPTION:
Cross-sectional prospective analysis of clinical efectiveness of a diabetes educational program to improve intermittently continuous glucose monitoring (iCGM) adherence in adult type 1 diabetes (T1D) patients. Glycometric data obtained through deidentified downloads from isCGM´s webpage. Primary outcome was time in range (TIR) 3.0-10 mmol/L (70-180 mg/d) change after the heatwave. Data analysis is conducted using SPSS (Chicago, IL) statistics software. Results are presented as mean ± SD values or percentages. A paired Student's t-test or a Wilcoxon signed-rank test were used for the analysis of differences. Comparisons between proportions were analyzed using a chi-squared test. A P value < 0.05 was considered statistically significant. The protocol was approved by the reference Castilla-La Mancha Public Health Institute Ethic Committee (C-558).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Flash user for at least 6 months.
* Treatment with multiple daily insulin injections (MDI).
* Daily scan Flash frequency 4 or less

Exclusion Criteria:

* Other types of diabetes
* Other types of diabetes treatment different from MDI (pe insulin pump)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Adherence to Flash 1 | 14 days
  Number of intermittently scanned continuous glucose monitoring daily scanning (number of scans per day)

SECONDARY OUTCOMES:
Time in range | 14 days
  Time in range (TIR) 3.0-10 mmol/L (70-180 mg/d) of interstitial glucose
Adherence to Flash 2 | 14 days
  Time of use of intermittently scanned continuous glucose monitoring (% possible time of use)
Time below range 1 (TBR1) | 14 days
  Time bellow range <3.9 mmol/L (<70 mg/dL) of the interstitial glucose
Time below range 2 (TBR2) | 14 days
  Time bellow range <3 mmol/L (<54 mg/dL) of the interstitial glucose
Time above range 1 (TAR1) | 14 days
  Time above range >10 mmol/L(>180 mg/dL) of the interstitial glucose
Time above range 2 (TAR2) | 14 days
  Time above range >13.9 mmol/L (>250 mg/dL) of the interstitial glucose
Coefficient of variation percentage (CV) | 14 days
  Coefficient of variation percentage of interstitial glucose
Glucose management index | 14 days
  Glucose management index of interstitial glucose
Time in hypoglycemia | 14 days
  Daily time in hypoglycemia (<3.9 mmol/L, <70 mg/dL) of interstitical glucose
Hypoglycemia frequency | 14 days
  Number of daily hypoglycemic events (<3.9 mmol/L, <70 mg/dL) of interstitical glucose
Percentage of patients attaining the the International Consensus on Time in Range (ICTR) | 14 days
  Percentage of patients (from total) attaining TIR>70%, TBR1<4%, TBR2<1%, TAR1<25%, TAR2<5% and CV <36%

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Moreno-Fernandez, PhD, Principal Investigator — Ciudad Real General University Hospital
Locations (1):
- Ciudad Real General University Hospital, Ciudad Real, Spain

IPD SHARING:
Plan to Share IPD: Yes
Under other researchers request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available after 1 month of the request and for a 3-month period.
Access Criteria: After request study from IP and ethic comittee.

REFERENCES:
- [Result] Chatterjee S, Davies MJ, Heller S, Speight J, Snoek FJ, Khunti K. Diabetes structured self-management education programmes: a narrative review and current innovations. Lancet Diabetes Endocrinol. 2018 Feb;6(2):130-142. doi: 10.1016/S2213-8587(17)30239-5. Epub 2017 Sep 29. PMID 28970034
- [Result] Hermanns N, Ehrmann D, Schipfer M, Kroger J, Haak T, Kulzer B. The impact of a structured education and treatment programme (FLASH) for people with diabetes using a flash sensor-based glucose monitoring system: Results of a randomized controlled trial. Diabetes Res Clin Pract. 2019 Apr;150:111-121. doi: 10.1016/j.diabres.2019.03.003. Epub 2019 Mar 4. PMID 30844467
- [Result] Bolinder J, Antuna R, Geelhoed-Duijvestijn P, Kroger J, Weitgasser R. Novel glucose-sensing technology and hypoglycaemia in type 1 diabetes: a multicentre, non-masked, randomised controlled trial. Lancet. 2016 Nov 5;388(10057):2254-2263. doi: 10.1016/S0140-6736(16)31535-5. Epub 2016 Sep 12. PMID 27634581
- [Result] Dunn TC, Xu Y, Hayter G, Ajjan RA. Real-world flash glucose monitoring patterns and associations between self-monitoring frequency and glycaemic measures: A European analysis of over 60 million glucose tests. Diabetes Res Clin Pract. 2018 Mar;137:37-46. doi: 10.1016/j.diabres.2017.12.015. Epub 2017 Dec 24. PMID 29278709
- [Result] Gomez-Peralta F, Dunn T, Landuyt K, Xu Y, Merino-Torres JF. Flash glucose monitoring reduces glycemic variability and hypoglycemia: real-world data from Spain. BMJ Open Diabetes Res Care. 2020 Mar;8(1):e001052. doi: 10.1136/bmjdrc-2019-001052. PMID 32198165